CLINICAL TRIAL: NCT06322732
Title: Optimization of Routine Obstetric and Neonatal Care in the Management of Severe Perinatal Asphyxia in Term or Near-term Newborns: Analysis of Sub-optimal Care
Acronym: OptiNeoCare
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP191125
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Perinatal Asphyxia
Keywords: Hypoxic-ischemic encephalopathy; perinatal asphyxia; neonatal death; suboptimal care; confidential inquiry
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Perinatal Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newborn at or near term: Newborn at or near term (≥ 36 weeks of amenorrhea), considered to be alive at the onset of labor and presenting severe perinatal asphyxia

SUMMARY:
The purpose of this study is to identify and analyze suboptimal perinatal (obstetric-pediatric) care in the occurrence and management of severe perinatal asphyxia or death of the newborn at or near term.

Perinatal asphyxia is a serious and often unexpected pathology, requiring urgent multidisciplinary care (obstetric - pediatric - intensive care, etc.) with a high level of technical expertise and care coordination. Because of its rarity and complexity, it may be subject to suboptimal care.

The aim of this study is to provide feedback within the center itself, coupled in 1/3 of cases with a confidential investigation into the search for and understanding of suboptimal care.

Primary endpoint:

Frequency of optimal or non-optimal maternal and neonatal management of hypoxic-ischemic encephalopathy (AIE) or neonatal death related to severe perinatal asphyxia.

DETAILED DESCRIPTION:
Perinatal asphyxia at term is a severe pathology that can lead to peripartum death or a birth in vital distress with neurological damage known as anoxic-ischemic encephalopathy (AIE), representing 1.6 per thousand births. In this unexpected and urgent situation, obstetric and neonatal management will have a decisive impact on the neonatal and neurological prognosis of the newborn. Despite a significant improvement in prognosis in recent years, it remains severe, with an estimated risk of death of 15-20% and moderate to severe disability in survivors of 30%.

The management of severe perinatal asphyxia combines a large number of risks that have been identified as providing suboptimal care in a patient deemed to be vulnerable. Batlle showed in an obstetrical clinical audit, in the form of a peer review in France in 2010, that half the cases of per-partum asphyxia audited were considered "possibly or certainly avoidable". Similar results were found in studies in Denmark and Sweden. Chevallier et al in France showed that around 35% of newborns requiring hypothermia did not receive it in accordance with French recommendations. The aim of analyzing this sub-optimal care is to identify the systematic factors that led to the error, and to suggest solutions to avoid similar cases in the future.

Corrective action has been taken on the basis of these studies: "Every case of asphyxia could be used as an example for learning" is the title of an article proposing recommendations for obstetric clinical practice based on audits of perinatal asphyxia cases. In Queensland, the implementation of a national education program on fetal heart rate reading has led to a significant reduction in the incidence of AIS from 250 to 160 events/100,000 live births. In the UK, a pragmatic approach has been initiated to improve prognosis in the context of perinatal asphyxia. "Each Baby Count" https://www.rcog.org.uk/eachbabycounts, is a national platform recording every case of perinatal asphyxia and AIE, and collecting data on sub-optimal care. This work will help to improve the quality of care both locally and nationally.

These experiences suggest that the identification of sub-optimal obstetric and neonatal care through a voluntary approach by the centers can lead to improved prevention and management. In France, serious adverse events are analyzed during morbidity and mortality reviews, which remain internal to the facilities and have limited impact at national level. The aim of this study is to describe cases of death or HIE, to analyze the risk factors and to assess the optimality of care in both obstetrics and pediatrics.

ELIGIBILITY:
Inclusion Criteria:

- Newborn at or near term (≥ 36 weeks of amenorrhea), considered to be alive at the onset of labor and presenting severe perinatal asphyxia

Severe perinatal asphyxia is considered if

1. Severity in its impact on the newborn:

   • a neonatal death during the initial hospitalization, since birth and before a possible return home, before D28 ".

   OR
   * moderate to severe anoxic-ischemic encephalopathy OR
   * a newborn hospitalized in the first week of life for hypoxic-ischemic encephalopathy or convulsions related to a perpartum event.

   AND
2. Biological perinatal asphyxia:

   * a pH (arterial or, failing that, venous) ≤ 7.10 or base deficit ≥ 16mmol/L or lactates ≥ 11mmol/L during the first three hours of life OR
   * In the absence of biological documentation of metabolic acidosis, an Apgar ≤ 5 to 5 minutes of life or the need for neonatal resuscitation (ventilatory support at birth and Apgar score ≤ 7 to 10 minutes of life).
   * If none of the biological elements are available in the file, keep the clinical inclusion criteria below (In the absence of biological and clinical Apgar data (home delivery type), inclusion may be based on neonatal outcome (death - hypoxic ischemic encephalopathy - neonatal convulsions).

Exclusion Criteria

* Fetal death in utero prior to hospital admission
* Medical termination of pregnancy
* Severe malformations with potential impact on child survival and development.
* Neonatal encephalopathy not due to perinatal asphyxia

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cases of severe perinatal asphyxia will be drawn from the general population of full-term or near-term deliveries in the participating network's maternity units, whether public, private or home birth, and for all types of maternity unit (type 1 - 2 or 3)
Sampling Method: Non-Probability Sample
Enrollment: 336 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
sub-optimal perinatal care | 1 year
  Identify and analyze sub-optimal perinatal (obstetric-pediatric) care in the occurrence and management of severe perinatal asphyxia or death of the newborn at or near term.

SECONDARY OUTCOMES:
Frequency of suboptimal care | 1 year
  Describe the frequency and context of HIE or neonatal death secondary to severe perinatal asphyxia.
Relationship | 1 year
  Evaluate possible relationships between suboptimal care and the occurrence of severe perinatal asphyxia
Outcome | 1 year
  Evaluate possible relationships between suboptimal care and the outcome of newborns in terms of mortality and neurological morbidity
Characteristics of suboptimal care | 1 year
  Analyze the characteristics of sub-optimal care identified by experts
Determinantes of suboptimal care | 1 year
  Assessing the determinants of suboptimal care
Ad-hoc survey | 1 year
  Evaluate the relevance of an ad-hoc survey versus a confidential survey on the analysis of sub-optimal care.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle GUELLEC-RENNE, MD, PhD, Study Director — Intensive care unit - L'archet University Hospital of Nice Côte d'Azur; Gilles KAYEM, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Yes
Undecided

REFERENCES:
- [Derived] Guellec I, Ancel PY, Abdoul H, Garabedian C, Verspyck E, Huissoud C, Delnaud M, Graesslin B, Desplanches T, Cambonie G, Tourneux P, Debillon T, Mitha A, Loron G, Favrais G, Badr M, Chapeliere S, Brasseur-Daudruy M, Gonzalez Estevez M, Rigouzzo A, Delorme P, Kayem G. OptiNeoCare: optimisation of routine care in the management of severe perinatal asphyxia in full-term or near-term newborns - study protocol for analysis of suboptimal care by confidential inquiries and e-self report. BMJ Open. 2025 Jul 5;15(7):e106093. doi: 10.1136/bmjopen-2025-106093. PMID 40617609